CLINICAL TRIAL: NCT05885997
Title: Implementing a Home Blood Pressure Monitoring Program to Improve Hypertension Control in a Primary Care Network: the MonitorBP Cluster Randomized Trial
Brief Title: Implementing a Home Blood Pressure Monitoring Program in Primary Care
Acronym: MonitorBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Weill Medical College of Cornell University (Other); New York Presbyterian Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ian Kronish, Associate Professor of Medicine at CUIMC, Associate Director of the Center for Behavioral Cardiovascular Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAS5544; R01HL152699 (NIH)
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: home blood pressure monitoring; remote patient monitoring; self-measured blood pressure monitoring; implementation science
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be blinded to group assignment when analyzing electronic health record data to determine the effectiveness of the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention Clinics, Pre-Implementation Period (Experimental): Usual care
  Interventions: Other: Usual care
- Intervention Clinics, Post-Implementation Period (Experimental): Access to Supported HBPM program plus a multifaceted implementation strategy designed to increase uptake of the program by primary care patients with uncontrolled hypertension
  Interventions: Behavioral: Supported HBPM program plus multifaceted implementation strategy
- Control Clinics, Pre-Implementation Period (Other): Usual care
  Interventions: Other: Usual care
- Control Clinics, Post-Implementation Period (Other): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Supported HBPM program plus multifaceted implementation strategy — Supported HBPM Program:
  * Patients are loaned a wireless home BP device or use their own device
  * Navigator or app support for onboarding and engaging patients in HBPM
  * Nursing or app support for monitoring and triaging home BP data for extreme readings
  * EHR integration of order for program and home BP data, with weekly feedback of home BP results to clinicians within the EHR
  Multifaceted implementation strategy:
  * Clinician education about the benefits of the program as well as training in how to refer and manage patients who are enrolled
  * Prompts and reminders to increase clinician referrals
  * Instructional materials for patients and clinicians
  * Problem-solving meetings to tailor implementation for individual practices
  Arms: Intervention Clinics, Post-Implementation Period
Other: Usual care — Usual care
  Arms: Control Clinics, Post-Implementation Period; Control Clinics, Pre-Implementation Period; Intervention Clinics, Pre-Implementation Period

SUMMARY:
The goal of this research is to determine whether a theory-informed implementation strategy is successful at increasing the uptake of a supported home blood pressure monitoring (HBPM) program as well as to determine the effectiveness of this evidence-based practice when implemented across multiple practices serving a diverse patient population.

DETAILED DESCRIPTION:
Hypertension guidelines now strongly recommend that patients with hypertension monitor their blood pressure (BP) at home (i.e., home BP monitoring; HBPM) as an approach to improving BP control so long as HBPM is conducted with clinical support (i.e., supported HBPM). Yet, few health systems have systematically implemented HBPM programs, and less than 20% of hypertensive patients routinely measure their BP at home, resulting in a gap in the translation of evidence-based recommendations into practice.

While there is strong evidence for Supported HBPM from pragmatic randomized controlled trials (RCTs), the evidence has been generated from the subgroup of patients and clinicians who volunteered to participate in trials, and the sample sizes have been in the hundreds of patients. There remains a gap in assessing the effectiveness of a scaled-up HBPM program that seeks to maximize the enrollment of primary care patients with uncontrolled hypertension.

Accordingly, in partnership with health system leaders at New York-Presbyterian Hospital (NYP), Columbia University Irving Medical Center, and Weill Cornell Medicine, the study investigator leveraged a system-wide investment in telemedicine to develop a telemonitoring-enabled Supported HBPM program. The Supported HBPM program consists of two options for obtaining electronic health record (EHR)-integrated home BP data. The low resource intensity option is designed for patients that can obtain valid home BP devices and are comfortable using the patient portal. It includes digital support to prompt patients to track their home BP readings in the patient portal using their own BP devices with automated triage support for extreme readings. The high resource intensity option is designed for patients that need additional support with HBPM. It involves navigator support with obtaining and using loaned home BP devices that wirelessly transmit data into the EHR and nursing support to triage extreme readings. Both programs can be ordered by clinicians in the EHR and both provide clinicians with weekly summaries of home BP readings with average home BP already calculated.

The study investigator concurrently followed a theory-driven process (the Behavior Change Wheel) to develop an implementation strategy aimed at increasing uptake of the Supported HBPM program. The study investigator now plans to implement and evaluate the Supported HBPM program across practices in the NYP, Weill Cornell Medicine, and ColumbiaDoctors primary care network which is comprised of a socioeconomically diverse patient population.

The study will evaluate the program by conducting a parallel-group cluster randomized trial in which 15 practices will be matched and then randomly assigned to early implementation of the Supported HBPM program (intervention) versus usual care with delayed implementation (i.e., wait-list control). Data will be retrospectively collected from a 12 month period before implementation (pre-implementation periods) as well as from a 12 month period after implementation (post-implementation period) to assess outcomes.

If successful, this project will provide a roadmap for widely implementing an EHR-integrated Supported HBPM program, and will accelerate a change in the paradigm of hypertension management from the office to the home.

ELIGIBILITY:
Patient-level

Inclusion Criteria:

* Hypertension (as per International Statistical Classification of Diseases and Related Health Problems (ICD)-10 codes)
* At least one completed primary care office visit during relevant 6-month pre implementation or post-implementation study time period
* Age 18-85 years old

Exclusion Criteria:

* Advanced dementia or other measure of frailty (as per ICD-10 codes)
* Pregnancy during measurement period (as per ICD-10 codes)
* Stage 5 or end-stage kidney disease (as per ICD-10 codes)
* Terminal illness/in hospice care (as per ICD-10 codes)

Practice-level

Inclusion Criteria:

* Primary care practice that provides care to adult patients affiliated with New York Presbyterian's Ambulatory Care Network, ColumbiaDoctors, or Weill Cornell Medicine, including practices that specialize in HIV medicine

Exclusion Criteria:

* Medical director declines participation in the trial
* Site for pilot testing the supported HBPM program or its implementation strategy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23928 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient's office systolic blood pressure (SBP) | 12 months
  Change in patient's office systolic blood pressure (SBP) from index visit to last visit during the subsequent 12 months, among patients with uncontrolled hypertension at the index visit

SECONDARY OUTCOMES:
Office diastolic blood pressure (DBP) | 12 months
  Change in patient's office diastolic blood pressure (DBP) from index visit to last visit during the subsequent 12 months, among patients with uncontrolled hypertension at the index visit
Change in patient's antihypertensive medication regimen intensity | 12 months
  Change in patient's antihypertensive medication regimen intensity as calculated by the Therapeutic Intensity Score from index visit to last visit during the subsequent 12 months, among patients with uncontrolled hypertension at the index visit
Antihypertensive medication adherence | 12 months
  Change in the proportion of days covered by antihypertensive medications from the 6 months prior to the index visit to the last 6 months of the 12-month follow-up period, among patients with uncontrolled hypertension at the index visit. Antihypertensive medication adherence will be calculated for each prescribed class of medication and then averaged across all classes.
Uncontrolled hypertension | 12 months
  Percentage of patients whose last office BP during the 12-month follow-up period was SBP>= 140 mmHg or DBP >= 90 mmHg, among all eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Ian Kronish, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data archive that contains raw study data will be posted on an open science platform.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of major study activities.
Access Criteria: Access to the data archive will be provided upon request